CLINICAL TRIAL: NCT00003617
Title: Protocol for a Randomised Trial of Observation Versus Chlorambucil After Anti-Helicobacter Therapy in Low Grade Gastric Lymphoma
Brief Title: Chlorambucil Compared With No Further Therapy Following Anti-Helicobacter Therapy in Treating Patients With Low-Grade Lymphoma of the Stomach
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lymphoma Trials Office (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066695; BNLI-LY03; EU-98040
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-04

CONDITIONS: Gastric Cancer
Keywords: stage I gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chlorambucil; Clarithromycin; Omeprazole; Tinidazole

INTERVENTIONS:
Drug: chlorambucil
Drug: clarithromycin
Drug: omeprazole
Drug: tinidazole

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known whether chlorambucil is more effective than observation in treating low-grade lymphoma of the stomach.

PURPOSE: Randomized phase III trial to compare the effectiveness of chlorambucil with that of no further therapy following anti-Helicobacter therapy in treating patients with low-grade lymphoma of the stomach.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy and response rate of triple antibiotic therapy for Helicobacter pylori in the healing of lesions in patients with low grade gastric lymphoma. II. Assess the efficacy of chlorambucil in the prevention of relapse in patients after complete eradication of low grade gastric lymphoma. III. Determine the natural history of unresected or partially resected low grade gastric lymphoma treated medically.

OUTLINE: This is a randomized study. Patients are randomized to receive chlorambucil or placebo. Patients receive omeprazole daily for 1 week. Clarithromycin and tinidazole are administered twice daily for 1 week for the eradication of H. pylori infection. Patients are assessed every 2-3 months by endoscopy. Patients may receive a maximum of 3 courses of treatment every 2-3 months. Other regimens may be used if full eradication of H. pylori is not achieved. Patients who achieve complete response (eradication of H. pylori) are randomized to receive oral chlorambucil or placebo daily for 14 days. Treatment is repeated every 28 days for 6 courses. Patients are followed every 6 months for 2 years, then yearly thereafter.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Endoscopically diagnosed, unresected, partially resected, or completely resected low grade (stage I) gastric lymphoma Prior diagnosis of H. pylori infection No nodal metastases Microbiological evidence of current H. pylori infection required No pathological evidence of enlarged abdominal lymph nodes by CT scan Gastroscopic ultrasound evidence of enlarged nodes allowed, if CT scan normal

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1995-03

CONTACTS AND LOCATIONS:
Overall Officials: Barry W. Hancock, MD, Study Chair — Cancer Research Centre at Weston Park Hospital
Locations (30):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Oncology Centre Institute, Warsaw, Poland
- Frere Hospital, Central Region, South Africa
- Ospedale San Giovanni, Bellinzona, Switzerland
- United Kingdom (26):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Royal Free Hospital, Hampstead, London, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Leeds Teaching Hospital Trust, Leeds, England
  - Charing Cross Hospital, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Salford Royal Hospitals NHS Trust, Salford, England
  - Weston Park Hospital, Sheffield, England
  - Royal Marsden Hospital, Sutton, England
  - Good Hope Hospital Trust, West Midlands, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - York District Hospital, York, England
  - Kettering General Hosptial, Kettering, Northants
  - James Paget Hospital, Norfolk
  - Rotherham District General Hospital-NHS Trust, Rotherham
  - Salisbury District Hospital, Salisbury
  - Staffordshire General Hospital, Stafford

REFERENCES:
- [Result] Hancock BW, Qian W, Linch D, Delchier JC, Smith P, Jakupovic I, Burton C, Souhami R, Wotherspoon A, Copie-Bergman C, Capella C, Traulle C, Levy M, Cortelazzo S, Ferreri AJ, Ambrosetti A, Pinotti G, Martinelli G, Vitolo U, Cavalli F, Gisselbrecht C, Zucca E. Chlorambucil versus observation after anti-Helicobacter therapy in gastric MALT lymphomas: results of the international randomised LY03 trial. Br J Haematol. 2009 Feb;144(3):367-75. doi: 10.1111/j.1365-2141.2008.07486.x. Epub 2008 Nov 22. PMID 19036078
- [Result] Bertoni F, Conconi A, Capella C, Motta T, Giardini R, Ponzoni M, Pedrinis E, Novero D, Rinaldi P, Cazzaniga G, Biondi A, Wotherspoon A, Hancock BW, Smith P, Souhami R, Cotter FE, Cavalli F, Zucca E; International Extranodal Lymphoma Study Group; United Kingdom Lymphoma Group. Molecular follow-up in gastric mucosa-associated lymphoid tissue lymphomas: early analysis of the LY03 cooperative trial. Blood. 2002 Apr 1;99(7):2541-4. doi: 10.1182/blood.v99.7.2541. PMID 11895791
- [Result] Zucca E, Roggero E, Delchier J, et al.: Interim evaluation of gastric malt lymphoma response to antibiotics in the ongoing LY03 randomized cooperative trial of observation vs chlorambucil after anti-helicobacter therapy. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A12, 2000.